CLINICAL TRIAL: NCT03303521
Title: A Phase 3b, Multicenter, Prospective, Randomized, Double Blind, Placebocontrolled Study to Reduce Incidence of Pre-dialysis Hyperkalemia With Sodium Zirconium Cyclosilicate (DIALIZE)
Brief Title: A Study to Test Whether ZS (Sodium Zirconium Cyclosilicate) Can Reduce the Incidence of Increased Blood Potassium Levels Among Dialized Patients.
Acronym: DIALIZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9480C00006; 2017-003029-14 (EudraCT Number)
Record Dates: First submitted 2017-09-26; First posted 2017-10-06 (Actual); Results first posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Zirconium Cyclosilicate (ZS) (Experimental): Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of ZS 5g depending on dose level assigned to a patient per non-dialysis days.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS)
- Placebo (Placebo Comparator): Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) Single dose contains from 1 to 3 sachets of Placebo depending on dose level assigned to a patient per non-dialysis days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) .
  Single dose contains from 1 to 3 sachets of Placebo depending on dose level assigned to a patient per non-dialysis days.
  Arms: Placebo
Drug: Sodium Zirconium Cyclosilicate (ZS) — Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose) .
  Single dose contains from 1 to 3 sachets of ZS 5g depending on dose level assigned to a patient per non-dialysis days.
  Arms: Sodium Zirconium Cyclosilicate (ZS)

SUMMARY:
The purpose of this study is to evaluate the efficacy of ZS in the treatment of hyperkalemia in patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged ≥ 18 years at screening Visit 1. For patients aged <20 years and enrolled in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative.
3. Receiving hemodialysis (or hemodiafiltration) 3 times a week for treatment of endstage renal disease (ESRD) for at least 3 months before randomization.
4. Patients must have hemodialysis access consisting of an arteriovenous fistula, AV graft, or tunneled (permanent) catheter which is expected to remain in place for the entire duration of the study.
5. Pre-dialysis serum K >5.4 mmol/L after long inter-dialytic interval and >5.0 mmol/L after one short inter-dialytic interval during screening (as assessed by central lab).
6. Prescribed dialysate K concentration ≤ 3 mmol/L during screening
7. Sustained Qb ≥200 ml/min and spKt/V ≥1.2 (or URR ≥ 63) on stable hemodialysis/hemodiafltration prescription during screening with prescription (time, dialyzer, blood flow [Qb], dialysate flow rate [Qd] and bicarbonate concentration) expected to remain unchanged during study
8. Heparin dose (if used) must be stable during screening and expected to be stable during the study
9. Subjects must be receiving dietary counseling appropriate for ESRD patients treated with hemodialysis/hemodiafiltration as per local guidelines, which includes dietary potassium restriction.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca, including ZS Pharma staff and/or staff at the study site)
2. Hemoglobin <9 g/dL on screening (as assessed on Visit 1)
3. Lack of compliance with hemodialysis prescription (both number and duration of treatments) during the two-week period preceding screening (100% compliance required)
4. Patients treated with sodium polystyrene sulfonate (SPS, Kayexalate, Resonium), calcium polystyrene sulfonate (CPS, Resonium calcium) or patiromer (Veltassa) within 7 days before screening or anticipated in requiring any of these agents during the study
5. Myocardial infarction, acute coronary syndrome, stroke, seizure or a thrombotic/thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism, but excluding vascular access thrombosis) within 12 weeks prior to randomization
6. Laboratory diagnosis of hypokalemia (K < 3.5 mmol/L), hypocalcemia (Ca < 8.2 mg/dL; for Japan hypocalcemia is defined as albumin-corrected Ca < 8.0 mg/dL), hypomagnesemia (Mg < 1.7 mg/dL) or severe acidosis (serum bicarbonate 16 mEq/L or less) in the 4 weeks preceding randomization
7. Pseudohyperkalemia secondary to hemolyzed blood specimen (this situation is not considered screening failure, sampling or full screening can be postponed to a later time as applicable).
8. Severe leukocytosis (>20× 10^9/L) or thrombocytosis (≥450 × 10^9/L) during screening
9. Polycythemia (Hb >14 g/dL) during screening
10. Diagnosis of rhabdomyolysis during the 4 weeks preceding randomization
11. Patients treated with lactulose, xifaxan (rifaximin) or other non-absorbed antibiotics for hyperammonemia within 7 days prior to the first dose of study drug
12. Patients unable to take oral ZS drug mix
13. Scheduled date for living donor kidney transplant
14. Patients with a life expectancy of less than 6 months
15. Female patients who are pregnant or breastfeeding
16. Females of childbearing potential, unless using contraception as detailed in the protocol or sexual abstinence.
17. Known hypersensitivity or previous anaphylaxis to ZS or to components thereof
18. Participation in another clinical study with an investigational product during the last 1 month before screening
19. Any medical condition, including active, clinically significant infection, that in the opinion of the investigator or Sponsor may pose a safety risk to a patient in this study, which may confound safety or efficacy assessment and jeopardize the quality of the data, or may interfere with study participation
20. Presence of cardiac arrhythmias or conduction defects that require immediate treatment
21. History of alcohol or drug abuse within 2 years prior to randomization
22. Previous randomization in the present study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — NSUH,Dept of Medicine,300 Community Drive,Manhasset,NY11030
Locations (47):
- United States (14):
  - Research Site, Los Angeles, California
  - Research Site, Ontario, California
  - Research Site, San Dimas, California
  - Research Site, Whittier, California
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Paterson, New Jersey
  - Research Site, Fresh Meadows, New York
  - Research Site, Great Neck, New York
  - Research Site, Ridgewood, New York
  - Research Site, The Bronx, New York
  - Research Site, East Providence, Rhode Island
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
- Japan (16):
  - Research Site, Hamamatsu
  - Research Site, Kumamoto
  - Research Site, Miyagi-gun
  - Research Site, Nagano
  - Research Site, Niigata
  - Research Site, Ora-gun
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sashima-gun
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Toride-shi
  - Research Site, Tsukuba
  - Research Site, Wakayama
  - Research Site, Yachiyo-shi
  - Research Site, Yokosuka-shi
- Russia (11):
  - Research Site, Kemerovo
  - Research Site, Kolomna
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Penza
  - Research Site, Podolsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- United Kingdom (6):
  - Research Site, Cardiff
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Swansea
  - Research Site, York

REFERENCES:
- [Derived] Fishbane S, Ford M, Fukagawa M, McCafferty K, Rastogi A, Spinowitz B, Staroselskiy K, Vishnevskiy K, Lisovskaja V, Al-Shurbaji A, Guzman N, Bhandari S. Potassium responses to sodium zirconium cyclosilicate in hyperkalemic hemodialysis patients: post-hoc analysis of DIALIZE. BMC Nephrol. 2022 Feb 8;23(1):59. doi: 10.1186/s12882-021-02569-7. PMID 35135481
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00006&attachmentIdentifier=c9e82fef-889a-4fa8-a7a4-d2f8c17e1653&fileName=D9480C00006_CSP_redacted.pdf&versionIdentifier=
- See also: D9480C00006 SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00006&attachmentIdentifier=bd3feeb6-4e7a-49da-8b34-b2ef1e35c582&fileName=D9480C00006_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Zirconium Cyclosilicate (SZC); Placebo: Suspension administered orally for a treatment period of eight weeks (4 weeks of dose adjustment, 4 weeks in stable dose).
  Single dose contains 1 to 3 sachets that should be suspended in 45 mL of water by patient and administered on non-dialysis days.
Period: Overall Study
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Started | 97 | 99
Completed | 92 | 96
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 0
Not completed — Kidney transplantation | 0 | 1
Not completed — Investigational product discontinuation | 0 | 1
Not completed — Transferred to non-study dialysis center | 1 | 0
Not completed — Non-comliance to study protocol | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo | Total
Number analyzed (Participants) | 97 | 99 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (13.84) | 60.4 (13.2) | 58.1 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 57 | 58 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 52 | 102
  Black Or African American | 11 | 8 | 19
  Asian | 33 | 33 | 66
  American Indian Or Alasa Native | 1 | 2 | 3
  Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: A subject was considered to be a responder if, during the evaluation period, they maintained a pre-dialysis serum potassium (S-K) between 4.0 and 5.0 mmol/L on at least 3 out of 4 dialysis treatments following the long inter-dialytic interval and did not receive rescue therapy. The S-K levels used for this analysis were based on the measurements obtained by the central laboratory.
Time Frame: Evaluation period runs over the last 4 weeks of the treatment period up to 8 weeks, starting after visit 11 and ending on visit 15, thus it comprises post-long inter-dialytic interval visits 12, 13, 14 and 15.
Population: Full Analysis Set (all randomized patients)
Measure: Number; unit: Percentage of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 97 | 99
Percentage of participants | 41.2 | 1.0
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 68.77, 95% CI 2-sided [10.85 to 2810.85]

2. Secondary Outcome: Percentage of Patients Needing Rescue Therapy
Description: Patients requiring any urgent intervention consistent with local practice patterns to reduce serum potassium (S-K) including insulin/glucose, beta-adrenergic agonists, sodium bicarbonate, K binders or any form of renal replacement therapy.
Time Frame: An 8 week overall treatment period (a 4 week adjustment phase plus a 4 week evaluation phase) and a 2 week follow up period.
Population: Full Analysis Set (all randomized patients)
Measure: Number; unit: Percentage of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 97 | 99
Percentage of participants | 2.1 | 5.1

3. Primary Outcome: Percentage of Responders When Accounting for Missing Central Laboratory Serum Potassium Data
Description: The sensitivity analysis assessed the impact of subjects classified as non-responders due to missing serum potassium (S-K) data. Missing central lab (c-lab) pre-dialysis values were imputed using corresponding pre-dialysis i-STAT (a portable blood analyser) measurements. In addition, a "last observation carried forward" (LOCF) approach was utilized to further impute missing values of pre-dialysis S-K during the evaluation period. This technique will replace missing c-lab S-K values with the last available non-missing pre-dialysis LIDI observation recorded for that patient (and this could be a c-lab value or an imputed c-lab value). The Primary endpoint analysis was repeated on the imputed data.
Time Frame: as for outcome 1
Population: Full Analysis Set (all randomized patients)
Measure: Number; unit: Percentage of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 97 | 99
Percentage of participants | 42.3 | 2.0
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 35.51, 95% CI 2-sided [8.53 to 309.48]

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from time of randomization throughout the treatment period and including the follow-up period (until Visit 16 or the last patient visit in the study), up to 10 weeks (Day 71 +/- 3 days). SAEs will be recorded from the time of informed consent.
Description: Safety Analysis Set (All randomized subjects who received at least 1 dose of investigational product, SZC or placebo. N=96 for SZC, N=99 for Placebo). Subjects excluded from the Safety Analysis Set (n=1 for SZC, n=0 Placebo) did not receive treatment.
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/96 | 0/99
Serious Adverse Events (participants affected / at risk) | 7/96 | 8/99
Other Adverse Events (participants affected / at risk) | 7/96 | 11/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) (N=96) | Placebo (N=99)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) (N=96) | Placebo (N=99)
Nasopharyngitis (Infections and infestations) | 3 (4) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT03303521/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03303521/SAP_001.pdf